CLINICAL TRIAL: NCT05836818
Title: PROmotion of FLU Vaccine Uptake in the Emergency Department - PROFLUVAXED
Acronym: PROFLUVAXED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Duke University (Other); Thomas Jefferson University (Other); University of Washington (Other); Baylor College of Medicine (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 21-34004B; R01AI166967-01 (NIH)
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Results first posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Influenza Vaccination
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: A three-arm cluster randomized control trial to determine the effect of vaccine messaging and a question about acceptance, a question about acceptance without messaging, and standard care affect vaccine uptake in the ED.
Who Masked: Outcomes Assessor
Masking Description: outcomes assessor will not know arm assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Question (Q) (Experimental): Subjects receive no vaccine messaging, but are asked a question about whether they would accept a vaccine
  Interventions: Other: Question (Q)
- Messaging (M) (Experimental): Subjects receive vaccine messaging and are asked a question about whether they would accept a vaccine
  Interventions: Other: Question (Q); Other: Messaging (M)
- Non intervention (No Intervention): Usual care

INTERVENTIONS:
Other: Question (Q) — Flu vaccine acceptance question: a question asked of participants about their willingness to accept a flu vaccine
  Arms: Messaging (M); Question (Q)
Other: Messaging (M) — Flu vaccine educational materials -videos and flyers containing flu vaccine educational information
  Arms: Messaging (M)

SUMMARY:
The goal of this research is to increase influenza vaccine acceptance and uptake in vulnerable populations whose primary (and often only) health care access occurs in emergency departments (ED Usual Source of Care Patients). Toward this goal, the investigators will conduct one on one interviews and focus groups with ED Usual Source of Care Patients and community partners and produce trusted messaging informational platforms (PROmotion of FLU VA(X)ccination in the Emergency Department - PROFLUVAXED) that will address barriers to flu vaccination, especially vaccine hesitancy. The investigators will then conduct a cluster-randomized, controlled trial of PROFLUVAXED platforms in six EDs to determine whether their implementation is associated with greater flu vaccine acceptance and uptake in ED Usual Source of Care Patients.

DETAILED DESCRIPTION:
Specific Aim I: To determine whether implementation of influenza vaccine trusted messaging platforms is associated with increased influenza vaccine uptake in unvaccinated ED patients.

At six EDs (Zuckerberg San Francisco General, UCSF Parnassus Medical Center [San Francisco, CA], Thomas Jefferson University Hospital [Philadelphia, PA], Ben Taub Hospital [Houston, TX], Harborview Medical Center [Seattle, WA], and Duke University Medical Center [Durham, NC]), investigators will conduct a cluster-randomized controlled trial of implementation of PROFLUVAXED trusted messaging platforms, with influenza vaccine uptake in the ED as the primary outcome. Hypothesis: Implementation of PROFLUVAXED trusted messaging platforms in EDs will be associated with increased influenza vaccine uptake in unvaccinated ED patients.

Specific Aim II: To determine whether implementation of influenza vaccine trusted messaging platforms in EDs is associated with increased influenza vaccine acceptance in unvaccinated ED patients. For this specific aim influenza vaccine acceptance in the ED assessed via ED survey will be the primary outcome. Hypothesis: Implementation of PROFLUVAXED trusted messaging platforms in EDs will be associated with increased influenza vaccine acceptance in unvaccinated ED patients.

Specific Aim III: To determine whether implementation of a protocol in which ED patients are asked whether they will accept an influenza vaccine in the ED (and notifying ED providers when they say they will accept it) is associated with increased influenza vaccine uptake in unvaccinated ED patients. Hypothesis: Implementation of an ED protocol in which patients are asked whether they will accept an influenza vaccine (and notifying ED providers when they say they will accept it) will be associated with increased influenza vaccine uptake in unvaccinated ED patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adults
2. Presenting to ED
3. Not already vaccinated for influenza in the current year
4. Able to provide informed consent
5. Fluent in English or Spanish
6. Anticipated ability to complete study intervention in ED i.e., able to watch a 3-minute videoclip

Exclusion Criteria:

1. Age < 18 years
2. Major trauma such that it will preclude survey
3. Inability to participate in a survey because of intoxication, altered mental status, or critical illness
4. Incarceration
5. Psychiatric hold
6. We will also exclude patients who state that they have already received an influenza vaccine and patients who are in the ED for suspected acute Covid or influenza illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 776 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Rodriguez, MD, Principal Investigator — University of California, San Francisco
Locations (8):
- United States (8):
  - San Francisco General Hospital Emergency Department, San Francisco, California
  - University of California San Francisco Parnassus, San Francisco, California
  - Duke University Hospital, Durham, North Carolina
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Jefferson Methodist Hospital, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Washington-Harborview Emergency Department, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodriguez RM, Eucker SA, Rafique Z, Nichol G, Molina MF, Kean E, O'Laughlin KN, Bezek SK, Goicochea K, Ford JS, Morse D, White J, Arreguin MI, Shughart L, Chavez CL, Glidden DV, Rising KL. Promotion of Influenza Vaccination in the Emergency Department. NEJM Evid. 2024 Apr;3(4):EVIDoa2300197. doi: 10.1056/EVIDoa2300197. Epub 2024 Mar 26. PMID 38776635

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Recruitment days across all sites
Period: Overall Study
Arm/Group | Question (Q) | Messaging (M) | Non Intervention
Started | 245; 270 Recruitment days across all sites | 214; 270 Recruitment days across all sites | 317; 270 Recruitment days across all sites
Completed | 244; 270 Recruitment days across all sites | 210; 270 Recruitment days across all sites | 313; 270 Recruitment days across all sites
Not Completed | 1; 0 Recruitment days across all sites | 4; 0 Recruitment days across all sites | 4; 0 Recruitment days across all sites
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Later found to be previously vaccinated | 0 | 1 | 3
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Allergic to vaccines | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Question (Q) | Messaging (M) | Non Intervention | Total
Number analyzed (Participants) | 244 | 210 | 313 | 767
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 49 [32 to 61] | 47 [33 to 59] | 44 [32 to 58] | 46 [32 to 59]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 104 | 99 | 150 | 353
  Male | 136 | 109 | 161 | 406
  Other | 4 | 2 | 2 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants could choose multiple answers and thus may be counted more than once
  Participants
    African American | 81 | 73 | 120 | 274
    American Indian/Alaska Native | 3 | 6 | 12 | 21
    Asian | 8 | 8 | 17 | 33
    Latinx | 50 | 52 | 56 | 158
    Native Hawaiian/Pacific Islander | 1 | 4 | 2 | 7
    Middle Eastern | 2 | 1 | 1 | 4
    White (Non-Latino) | 96 | 78 | 112 | 286
    Other | 20 | 14 | 24 | 58
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 244 | 210 | 313 | 767

OUTCOME MEASURES:

1. Primary Outcome: Influenza Vaccine Uptake at 30 Days Comparing Intervention M and Non Intervention
Description: Participant uptake of the influenza vaccine 30 days after enrollment assessed by confirmation of receipt of vaccine in one of 3 ways:
  1. Receipt in emergency department during index (enrollment) visit
  2. Electronic health record review 30 days after index visit
  3. Follow up phone call to participant at 30 days - We are asking patients if they received a flu vaccine since their index emergency department visit.
Time Frame: 30 days post index ED visit
Measure: Count of Participants; unit: Participants
Groups:
- Non Intervention: Usual care, no intervention given. Control group
Arm/Group | Messaging (M) | Non Intervention
Number analyzed (Participants) | 210 | 313
Participants | 86 | 47
Statistical Analysis 1: Comparison: Non Intervention; Adjusted difference 25.1 percentage points; Test type: Superiority; p < 0.0001, Regression, Logistic; Mixed effects logistic regression with a random center effect for within-center characteristics, and terms for calendar time and intervention; Adjusted difference = 25.1, 95% CI 2-sided [17 to 33.2]

2. Secondary Outcome: Vaccine Acceptance
Description: Participants who responded they would accept a vaccine of asked in the ED. Comparing Intervention M and Intervention Q groups
Time Frame: during ED visit
Measure: Count of Participants; unit: Participants
Arm/Group | Messaging (M) | Question (Q)
Number analyzed (Participants) | 210 | 244
Participants | 103 | 110

3. Secondary Outcome: Influenza Vaccine Uptake at 30 Days Comparing Intervention Q and Non-Intervention Group
Description: as for outcome 1
Time Frame: 30 days post index ED visit
Measure: Count of Participants; unit: Participants
Arm/Group | Question (Q) | Non Intervention
Number analyzed (Participants) | 244 | 313
Participants | 78 | 47

4. Other Pre Specified Outcome: Influenza Vaccine Uptake at 30 Days Comparing Intervention M and Intervention Q
Description: as for outcome 1
Time Frame: 30 days post index ED visit
Measure: Count of Participants; unit: Participants
Arm/Group | Messaging (M) | Question (Q)
Number analyzed (Participants) | 210 | 244
Participants | 86 | 78

ADVERSE EVENTS:
Time Frame: Up to 30 days post ED index visit
Arm/Group | Question (Q) | Messaging (M) | Non Intervention
All-Cause Mortality (participants affected / at risk) | 0/244 | 1/210 | 2/313
Serious Adverse Events (participants affected / at risk) | 0/244 | 0/210 | 0/313
Other Adverse Events (participants affected / at risk) | 0/244 | 0/210 | 0/313

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-03): https://cdn.clinicaltrials.gov/large-docs/18/NCT05836818/Prot_SAP_001.pdf
  • Informed Consent Form (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT05836818/ICF_002.pdf